CLINICAL TRIAL: NCT07283328
Title: Shaping Gut Microbiota Through a Dietary Intervention to Regulate Inflammatory Processes
Brief Title: Methionine Intake Microbiota
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Multiple Sclerosis Society of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 23.111
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: gut microbiota; methionine; diet intervention; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized interventional pilot study with cross-over intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methionine supplementation (Experimental): Methionine supplementation will be achieved using commercially available methionine supplement (content methionine 500 mg, trice daily) with a monography from Health Canada (NPN 80017685) and compared to placebo pills.
  Interventions: Behavioral: Methionine-restricted diet
- Placebo (Placebo Comparator): Consumption of placebo pill trice daily for 2 weeks
  Interventions: Behavioral: Methionine-restricted diet

INTERVENTIONS:
Behavioral: Methionine-restricted diet — Methionine-restricted diet (plant-based diet) is a feasible and palatable way to achieve 50% reduction in methionine intake. Reduction to around 800 mg/day methionine will be achieved using participants' selection from low-methionine plant-based and ready to eat meals for 100% of their meals, for 6 weeks. Participants will be provided with education and a list of low methionine content food (green) and high methionine (red) for eating out, snacks and homemade meals.

SUMMARY:
Pro-inflammatory immune cells play a pivotal role in multiple sclerosis, and the gut microbiota is increasingly recognized as a key factor shaping the immune system. This study aims to determine the impact of a dietary intervention (methionine-restricted diet-MR) on gut microbiota and inflammation in humans. A randomized interventional pilot study with cross-over intervention is conducted in 40 healthy participants. For all participants, the first two weeks (week 1+week 2) consist of baseline assessment on their usual diet, and week 3+week 4 consist of MR diet only. For group A, the week 5+week 6 are MR+1,500 mg daily supplementation of methionine and for group B are MR+placebo, with a cross-over for week 7+week 8. Usual diet is resumed for all participants during week 9+week 10. Gut microbiota, blood levels of methionine and its metabolites, as well as immune and inflammatory markers will be evaluated every 2 weeks. It is hypothesized that MR could be used in humans to prevent and alleviate the course of multiple sclerosis by shaping the gut microbiota towards an anti-inflammatory profile, and that the gut microbiota is a biomarker associated with successful dietary interventions targeting inflammation in multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* 20-50 years old
* On omnivorous/western diet
* Understanding French or English

Exclusion Criteria:

* B12 deficiency
* Glomerular filtration rate <75 ml/h
* Liver dysfunction
* Pregnant or lactating
* Active inflammatory or infectious disease
* Insulino-dependent diabetes
* Active cancer
* Eating disorder
* BMI < 18.5 kg/m2
* Severe food allergies or intestinal problems or active substance dependence that would prevent adherence to the experimental diet

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota | At the end of week 2, 4, 6, 8, 10.
  Lipocalin-2 will be measured in stools to assess for inflammation in the gut. Stool samples from a given participant (all timepoints) will be processed simultaneously for DNA extraction and sequencing. Amplification of hyper-variable regions V1-V3 of 16S with primers, 16S libraries preparation and sequencing (Génome Québec) will be performed. Microbiota diversity will be measured with Shannon and α-diversity indexes. To represent microbial communities' similarity/difference between groups, a principal coordinates analysis (PCoA) will be used. Data will be interpreted by using high dimensional class comparisons via linear discriminant analysis of effect size (LEfSe) and volcano plots to identify potential relationships between specific bacteria and immunological/metabolomics results and clinical data.

SECONDARY OUTCOMES:
Immune and inflammatory profile | At the end of week 2 ,4, 6, 8, 10.
  Established FACS panels will be used to characterize the complete immune profile including markers for B cells, T cells, myeloid cells, and CAMs implicated in gut and CNS homing. Validated multiplex immunoassays will be used on serum and supernatants to assess immune/inflammatory markers and metabolic markers (leptin, adiponectin, FGF21) in serum. In addition, sCD14, intestinal-type fatty acid-binding protein, and soluble suppression of tumorigenicity 2, which all correlated with gut damage in humans, will be measured.
Methionine level | At the end of week 2, 4, 6, 8, 10.
  Levels of methionine and its metabolites (SAM and SAH) will be measured by LC-MS (serum and PBMCs).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche du Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No